CLINICAL TRIAL: NCT06628440
Title: Development and Validation of a Mouth Assessment Tool for Orally Intubated Patients in Intensive Care Unit)
Acronym: MAT
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/48
Record Dates: First submitted 2024-08-27; First posted 2024-10-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Intensive Care
Keywords: intensive care; oral care; paramedical care; oro-tracheal intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: intensive care patient with oro-tracheal intubation
  Interventions: Other: oral condition assessment tool

INTERVENTIONS:
Other: oral condition assessment tool — Use of the Mat assessment tool by a nurse on the participant

SUMMARY:
Oro-tracheal Intubation uses oro-pharyngeal lesions, impacting on the length and quality of the patient's hospital stay.

There are no oral status assessment tools specifically adapted to orally intubated patients.

It is therefore necessary to create a new tool for assessing the condition of the oral cavity, specific to oro-intubated patients in intensive care.

The aim of the protocol is to evaluate the metrological performance of the newly-developed tool for assessing the state of the oral cavity in adult orally intubated intensive care patients.

DETAILED DESCRIPTION:
In France, according to the "medicalized information system program" national database, 230,000 adults are admitted to the intensive care unit every year, 40% of them undergoing invasive mechanical ventilation. That's 90,000 patients for whom an Oro-Tracheal Intubation (OTI) tube is inserted through the mouth into the trachea.

OTI causes oro-pharyngeal lesions, impacting on the length and quality of the patient's hospital stay.

As early as 48 hours after admission to intensive care, the patient's oral and dental condition deteriorates. Pressure lesions can occur, with the OTI probe responsible for 22% to 26% of pressure sores related to invasive equipment. Anarchic chewing also causes injuries to lips, tongue, gums, mucosa and teeth.

In time, these injuries can lead to swallowing disorders, a mechanism for feeding and protecting the airways, and impair the patient's quality of life.

Caregivers in intensive care units have developed mouth care protocols to maintain hygiene and comfort, and prevent lesions that can spread from the lips to the trachea during OTI.

Many mouth care protocols exist, but there is no "gold standard". Certain practices are encouraged as part of the prevention of Ventilator-Acquired Pneumonia (VAP) (mainly tooth brushing). Mouth care practices in France remain highly heterogeneous. In order to improve practices, it is essential not only to have best practice guidelines for preventing and treating lesions, but also to have appropriate and valid tools for assessing the oral condition of intubated patients. Good assessment is a prerequisite for good treatment/care.

To investigators knowledge, there are no oral status assessment tools specifically adapted to intubated patients.

Tools do exist for populations at risk due to age or chemotherapy, but these have often been created without multidisciplinary advice, validated in a population without OTI, and do not allow for an assessment of the state of the oral cavity appropriate to the problems of intubated patients.

It is therefore necessary to create a new tool for assessing the condition of the oral cavity, specific to oro-intubated patients in intensive care, by bringing together experts in intensive care, oral health, hygiene, wound healing and patient partners, and to validate it in this patient population. The tool must also be relevant to the fields of competence of nurses, for use in daily practice.

The aim of the protocol is to evaluate the metrological performance of the newly-developed tool for assessing the state of the oral cavity in adult oro-intubated intensive care patients.

ELIGIBILITY:
Inclusion Criteria:

* Person aged 18 or over
* Person hospitalized in an adult intensive care unit for medical, surgical, polyvalent or burns specialties.
* Person undergoing oro-tracheal intubation.
* Person affiliated with or benefiting from a social security scheme.
* Free and informed oral consent of the patient or his/her legal representative

Exclusion Criteria:

* Person undergoing Limitation or Cessation of Active Therapeutics
* Person wearing a multi-attachment fixed dental appliance (braces, multi-rings, brackets bonded to teeth)
* Person with oral damage making it impossible to measure one of the items on the oral cavity assessment tool (e.g.: removal of the tongue, etc.).
* Patient under protective supervision (safeguard of justice, curatorship, guardianship)
* Refusal of patient or legal representative to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in an adult intensive care undergoing oro-tracheal intubation.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Metrological performance of the Mouth Assessment Tool (MAT) | At inclusion (Day 0)
  The general evaluation criterion is the tool's metrological performance according to COSMIN (COnsensus-based Standards for the selection of health Measurement INstruments) psychometric criteria.

SECONDARY OUTCOMES:
Content validity of the Mouth Assessment Tool (MAT) | At inclusion (Day 0)
  Relevance of items, completeness of key concepts, understanding of items by target population
Construct validity of the Mouth Assessment Tool (MAT) | At inclusion (Day 0)
  Structural validity of the dimensional tool Hypothesis testing Measurement invariance in different population subgroups
Reliability of the Mouth Assessment Tool (MAT) | At inclusion (Day 0)
  Reproducibility Internal consistency

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU Angers, Angers
  - CHU de Bordeaux - Aile 1 Tripode, Bordeaux
  - CHU de Bordeaux - Aile 2 Tripode, Bordeaux
  - CHU de Bordeaux - Pellegrin, Bordeaux
  - CHU de Bordeaux - Saint André, Bordeaux
  - CHU Caen, Caen
  - CH Libourne, Libourne
  - CHU de Bordeaux - Haut Levêque, Pessac
  - Hôpital d'Instruction des Armées Sainte Anne, Toulon
  - Hôpitaux Nord Franche comté, Trévenans

IPD SHARING:
Plan to Share IPD: No